CLINICAL TRIAL: NCT05886283
Title: Qualitative and Quantitative Endothelium Changes After Cataract Surgery: Ultrasound Phacoemulsification vs Nanolaser Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Walid Zbiba, professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-03-2023
Record Dates: First submitted 2023-04-12; First posted 2023-06-02 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Effect of Cataract Surgery on Corneal Endothelium; About 2 Techniques
Keywords: cataract surgery; phacoemulsification; Nanosecond laser; endothelial cells density
MeSH Terms: interventions — Phacoemulsification

STUDY DESIGN:
Intervention Model Description: A randomized prospective, uncontrolled cohort study
Who Masked: Investigator
Masking Description: the investigator does not know the technique used to operate on the cataract during the follow-up
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound phaco groupe (Active Comparator): this group had US PHACO using the phaco-chop technique (Stellaris PC: Bausch + Lomb®)
  Interventions: Procedure: phacoemulsification; Procedure: utrasound phacoemulsification
- nanolaser phaco group (Active Comparator): this group underwent an NL PHACO (Cetus A.R.C. Laser system®)
  Interventions: Procedure: phacoemulsification; Procedure: nanolaser phacoemulsification

INTERVENTIONS:
Procedure: phacoemulsification — we started with a clear corneal incision of 2.2 mm at 9 o'clock and a port incision of 1 at 2 o'clock. Continuous Circular Capsulorhexis of 6 mm was performed under the same ophthalmic viscosurgical device. A hydro dissection was performed, then followed by phacoemulsification.
  the Nucleus has been treated using 2 different techniques After bimanual infusion/aspiration cortex removal and Visco expansion of the capsular bag, a hydrophobic single-piece: AcrySof acrylic IOL was implanted.
Procedure: utrasound phacoemulsification — US group:The nucleus was held with the phaco tip at a high vacuum. The phaco choppe was drawn towards the phaco tip to cleave it by a manual separation between the two instruments. The fragments were then aspirated with phaco power. The standard parameters used during phacoemulsification were a vacuum level of 500 mmHg, pressurized irrigation of 90 mmHg, and 40% of phaco power
  Arms: ultrasound phaco groupe
Procedure: nanolaser phacoemulsification — Laser group: The nucleus was fragmented using the shockwaves emanating from the phaco tip and then aspirated. The phaco chopper was used to accelerate the mechanical fragmentation of the nucleus and minimize the dissipated energy.
  Arms: nanolaser phaco group

SUMMARY:
Purpose: The aim of this study was to evaluate corneal endothelial cell density and morphology, central corneal thickness, and best visual acuity using US phacoemulsification or Nanosecond laser technique.

Setting: Department of ophthalmology, Nabeul, Tunisia. Design: Prospective cohort study. Methods: The study included eyes with nuclear cataract density grade 1, 2, 3, or 4 according to LOCS III, divided into two groups; Group 1 had conventional US, and group 2 had nanosecond laser. The Endothelial Cell Density (ECD), coefficient of variation (CoV) in cell size, percentage of hexagonal cells, central corneal thickness and best visual acuity were evaluated over 24 months.

DETAILED DESCRIPTION:
Methods:

A randomized prospective, uncontrolled cohort study was conducted at the Department of Ophthalmology of the Mohamed Taher Maamouri Hospital (MTMH) from March 2017 to May 2020. The MTMH ethics committee approved this study. All patients provided informed consent for the use of their data. The study adhered to all tenets of the declaration of Helsinki.

All patients underwent complete ocular examination including visual acuity, clinical corneal assessment, intraocular pressure (IOP) measurement, and nuclear hardness grading based on the lens opacity classification system III (LOCS III), commonly referred to in most studies. Only the nuclear component of the cataract (NO1 to NO4) was taken into account in the evaluation.

The endothelium of the central cornea was examined with a non-contact specular microscope (SM) (TOMEY CORP EM-4000).

Patients were randomly divided into 2 groups. Group 1 had US PHACO using the phaco-chop technique (Stellaris PC: Bausch + Lomb®) and group 2 underwent an NL PHACO (Cetus A.R.C. Laser system®).

The Cetus A.R.C. Laser system is composed of a base that generates a 4 to 5 ns pulsed Nd: YAG of 1064 nm wavelength laser with a pulse frequency up to 10 Hz and an optic fiber that transmits the laser pulses to the disposable single-use coaxial handpiece. The probe used has a total diameter of 720 µm, occupied in its center by a 320 µm quartz optical fiber that transferred the laser pulse towards a titanium plate in the phaco probe. The individual pulse energy ranged from 30 to 50 % of maximum power and the pulse frequency was 1-2 Hz.

The base unit is connected to the same phaco aspiration/irrigation system and is controlled by the pedal of that system.

In both groups, surgery started with a clear corneal incision of 2.2 mm at 9 o'clock and a port incision of 1 to 1.5 mm at 2 o'clock using the same knife. Continuous Circular Capsulorhexis (CCC) of 6 mm was performed under the same ophthalmic viscosurgical device (3% Sodium hyaluronate, 4% chondroitin sulfate, DuoVisc® Alcon ). A hydro dissection was performed, then followed by phacoemulsification.

In-group 1 (horizontal phaco chop): after cortex aspiration, the nucleus was held with the phaco tip at a high vacuum. The phaco chopper was then introduced from the side port incision to engage, under the lower edge of CCC. It was then drawn towards the phaco tip to cleave it by a manual separation between the two instruments. The same process continued for the two nuclear halves and the fragments were then aspirated with phaco power. The standard parameters used during phacoemulsification were a vacuum level of 500 mmHg, pressurized irrigation of 90 mmHg, and 40% of phaco power. Energy was expressed in % on the PHACO machine and initially converted into Watts according to the following curve "Figure 1" then into Joules based on the formula: Energy (Joules) = Power (Watts) × time (seconds).

In-group 2: The cortex and epinucleus were aspirated. The nucleus was fragmented using the shockwaves emanating from the phaco tip and then aspirated. The phaco chopper was used to accelerate the mechanical fragmentation of the nucleus and minimize the dissipated energy. The energy used was calculated automatically by the ARC Laser machine and was displayed on the screen.

In both groups, after bimanual infusion/aspiration cortex removal and Visco expansion of the capsular bag, a hydrophobic single-piece: AcrySof acrylic (SA60AT, Alcon) IOL was implanted. The duration of the whole procedure (in minutes) was noted.

Uncorrected Visual acuity (UVA) at 1 day postoperative and BCVA at 1 week, 1, 3, 6, and 24 months after surgery as well as corneal edema and anterior chamber (AC ) reaction were recorded. A visual outcome of 0.5 logarithm of the minimal angle of resolution (logMar) without correction was considered a successful result based on the World Health Organization definition (1, 15, 16). The SM was performed at 1 week, 1, 3, 6, and 24 months after surgery. The investigators reported endothelial cell density (EDC) (cell/ mm²), the percentage of hexagonal cells, coefficient of variation (CoV) in cell size, and central corneal thickness (CCT) at each follow-up visit.

All the data were analyzed using SPSS software (version 21.0; SPSS, Inc., Chicago, IL, USA). BCVA data was converted into log MAR for statistical analyses. Quantitative variables were presented as medians, means, and standard deviations. The investigators used Student's t-test for the independent series. Pearson's correlation coefficient was used for searching the statistical relationship or association between variables. A p-value < 0.05 was accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

-Senile cataract.

Non Inclusion Criteria:

* Preoperative endothelial cell count (ECC) less than 1500 cells/mm2.
* Pathological alterations of the anterior segment such as corneal opacities, cornea Guttata, uveitis, pseudoexfoliative syndrome, glaucoma, high myopia axil length (≥ 26 mm), or suffering from chronic pathologies that may affect corneal endothelium

Exclusion Criteria:

* Conversion from NL PHACO to US PHACO.
* Surgery was complicated with capsular rent and vitreous loss.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Endothelial cell density (ECD) | 2 years
  The endothelium of the central cornea was examined using a non-contact specular microscope (SM) (TOMEY CORP EM-4000).
Percentage of endothelial cell loss (ECL) | 2 years
  ECL was evaluated using a non-contact specular microscope (SM) (TOMEY CORP EM-4000).
Mean percentage of hexagonal cells | 2 years
  The mean percentage of hexagonal cells was evaluated using a non-contact specular microscope (SM) (TOMEY CORP EM-4000).
Mean coefficient of variance (CoV) | 2 years
  CoV was evaluated using a non-contact specular microscope (SM) (TOMEY CORP EM-4000).
Central corneal thickness (CCT) | 2 years
  CCT was evaluated using a non-contact specular microscope (SM) (TOMEY CORP EM-4000).
Uncorrected visual acuity (UVA) | 2 years
  UVA was evaluated at 1 day post-operatively
Best corrected visual acuity (BCVA) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Taher Maamouri Hospital, Nabeul, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zbiba W, Kharrat M, Sayadi S, Kallel Z, Marzouk G. Qualitative and quantitative endothelium changes after cataract surgery: ultrasound phacoemulsification vs. nanolaser technique. Front Med (Lausanne). 2023 Sep 21;10:1097404. doi: 10.3389/fmed.2023.1097404. eCollection 2023. PMID 37809334